CLINICAL TRIAL: NCT05532943
Title: A Seamless Phase I/IIa Clinical Study to Evaluate the Safety and Efficacy of Allogeneic Umbilical Cord Mesenchymal Stem Cells in Patients With Multiple Sclerosis
Brief Title: Evaluate the Safety and Efficacy of Allogeneic Umbilical Cord Mesenchymal Stem Cells in Patients With Multiple Sclerosis
Acronym: UMSC01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ever Supreme Bio Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ES-CMSC01-D1101
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- UMSC01 (Experimental): UMSC01 cells mixed with normal saline will be administered to patients after the onset of diagnosis of multiple sclerosis.
  Interventions: Biological: Allogeneic umbilical cord mesenchymal stem cells
- Placebo (Sham Comparator): For IV administration, normal saline will be administered to patients after the onset of diagnosis of multiple sclerosis. For IT administration, sham puncture procedure will partially penetrate without reaching subarachnoid space, and no spinal fluid will be drawn.
  Interventions: Biological: Control group

INTERVENTIONS:
Biological: Allogeneic umbilical cord mesenchymal stem cells — UMSC01 cells will be IV infusion followed by IT infusion with 12 months of follow up after treatment.
  Arms: UMSC01
Biological: Control group — Normal saline will be IV infusion followed by sham-IT infusion with 12 months of follow up after treatment.
  Arms: Placebo

SUMMARY:
This study is to identify the safety and efficacy of repeat IV(Intravenous) and IT(Intrathecal) administrations of UMSC01 in patients with MS. While anti-inflammatory drugs are routinely used for the treatment of MS by inhibiting immune responses, their effects on axon remyelination or neuroregeneration are limited. The combined systemic delivery of UCMSCs via intravenous injection and local administration of the cells by IT was to have safety and therapeutic efficacy for patients with MS.

DETAILED DESCRIPTION:
There is single arm in Phase I part: 6 patients will be enrolled sequentially for safety considerations. The patient will receive UMSC01 via IV followed by IT at day 28 as described in above. After all patients in Phase I complete the safety assessment by SMC without any major safety issue 4 weeks after the last UMSC01 administration, the Phase IIa part will be initiated. There are 2 arms in Phase IIa part: Sham-controlled with conventional treatment control and administration of UMSC01 with conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are willing to sign informed consent.
2. Male or female are age between 20 to 65 years old on date of consent.
3. Diagnosis of Relapsing-Remitting MS (RRMS) (≥1 clinically documented relapse in the past 12 months, ≥2 clinically documented relapses in the last 24 months or ≥ 1 gadolinium enhanced lesion or T2 new lesion in the last 12 months) or Secondary Progressive MS (SPMS) (EDSS increase ≥1.0 point (baseline EDSS ≤ 5.0) or ≥ 0.5 point (baseline EDSS ≥5.5), and ≥1 clinical relapse or ≥1 gadolinium enhanced lesion in the last 12 months)
4. MS diagnosis established between 2 to 15 years and EDSS score between 2.0 to 6.5 before enrollment
5. Patient has appropriated blood clotting function as assessed by the following laboratory requirements: PT, APTT ≤ 1.5X upper limit of normal (ULN).
6. Treatment failure (either ≥ 1 relapse, ≥ 1 new T2 lesion, ≥ one gadolinium enhanced lesion or EDSS deterioration) with at least one of MS disease modifying therapy as Interferon-β, Glatiramer acetate (Copaxone), Dimethyl fumarate (Tecfidera), Teriflunomide (Aubagio), Fingolimod (Gilenya), Ozanimod (Zeposia), Cladribine (Mavenclad), Siponimod (Mayzent), Ofatumumab (Kesimpta), or Natalizumab (Tysabri) for more than 6 months
7. All male patients and female patients with child-bearing potential (between puberty and 2 years after menopause) should use appropriate contraception method(s) for at least 4 weeks after UMSC01 treatment

Exclusion Criteria:

1. Pregnancy, lactation, and those who are not pregnant but did not, or unwilling to, take effective contraceptives measures 4 weeks before and after the treatment.
2. Patients with uncontrolled diabetes (fasting blood glucose > 250 mg/dL)
3. Patients with inadequate hepatic and renal function: AST and ALT > 5X ULN; eGFR < 30 mL/min.
4. Patients who are unable to undergo Brain MRI examination for any reason.
5. Patients who have medical history or current clinically active malignant tumor, peripheral neuropathy, myopathy or other clinically significant neurological diseases that will confound the evaluation of this study.
6. Patients who have immuno-compromised condition or is with known clinically significantly autoimmune conditions other than MS or is receiving immunosuppressive treatments other than MS treatment within 6 months.
7. With active infection that required systemic treatment
8. Patients who are participating in other clinical trials with an investigational product within 1 month.
9. Patients who were treated with cytotoxic medications during the last 1 month prior to the infusion.
10. Relapse of MS within1 month before UMSC01 infusion.
11. With anti-CD20 therapy, such as rituximab
12. Patients not suitable to participate the trial as judged by the Investigator(s)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint for Phase I portion | from visit 2 to 12-month follow-up period
  SAE, SUSAR, and AE incidences over the study period
Primary Endpoint for Phase IIa portion | from visit 2 to 12-month follow-up period
  CFB of EDSS to Visit 10

SECONDARY OUTCOMES:
Efficacy endpoint for phase I portion | from visit 2 to 12-month follow-up period
  CFB for EDSS of follow up visits (Visit 6-10)
Efficacy endpoint for phase I portion | from visit 2 to 12-month follow-up period
  CFB for brain MRI parameters of follow-up visits (Visit 6 -10)
Efficacy endpoint for phase I portion | from visit 2 to 12-month follow-up period
  Quality of life: CFB for MSQoL-54 questionnaire score of follow-up visits (Visit 6 -10)
Efficacy endpoint for phase I portion | from visit 2 to 12-month follow-up period
  CFB of T25FW scores of follow-up visits (Visit 6-10)
Efficacy endpoint for phase I portion | from visit 2 to 12-month follow-up period
  CFB of 9-HPT scores of follow-up visits (Visit 6-10)
Efficacy endpoint for phase I portion | from visit 2 to 12-month follow-up period
  CFB of PASAT scores of follow-up visits (Visit 6-10)
Efficacy endpoint for phase I portion | from visit 2 to 12-month follow-up period
  CFB of SDMT scores of follow-up visits (Visit 6-10)
Efficacy endpoint for phase I portion | from visit 2 to 12-month follow-up period
  CFB of RNFL thickness, measured by OCT of follow-up visits (Visit 6-10)
Efficacy endpoint for phase I portion | from visit 2 to 12-month follow-up period
  CFB of MSFC of follow-up visits (Visit 6-10)
Efficacy endpoints for phase IIa portion | from visit 2 to 6-month follow-up period
  Time to onset of CDW confirmed by EDSS at least 6 months
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  ARR (Annualized relapse rate), where relapse is defined as new or worsening neurological symptoms lasting for >24 hours
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  CFB of follow-up visits (Visit 6 -10) for EDSS
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  CFB of follow up visits (Visit 6-10) for brain MRI parameters
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  Quality of life: CFB of follow up visits (Visit 6-10) for MSQoL-54 questionnaire score
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  CFB of follow up visits (Visit 6-10) for T25FW scores
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  CFB of follow up visits (Visit 6-10) for 9-HPT scores
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  CFB of follow up visits (Visit 6-10) for PASAT scores
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  CFB of follow up visits (Visit 6-10) for SDMT scores
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  CFB of follow up visits (Visit 6-10) for RNFL thickness, measured by OCT
Efficacy endpoints for phase IIa portion | from visit 2 to 12-month follow-up period
  CFB of follow up visits (Visit 6-10) for MSFC
The safety endpoints are listed below for both phase I and IIa portions | from visit 2 to 12-month follow-up period
  SAE, SUSAR, and AE incidences over the study period
The safety endpoints are listed below for both phase I and IIa portions | from visit 2 to 12-month follow-up period
  CFB of laboratory data to subsequent visits
The safety endpoints are listed below for both phase I and IIa portions | from visit 2 to 12-month follow-up period
  CFB of physical examination to subsequent visits
The safety endpoints are listed below for both phase I and IIa portions | from visit 2 to 12-month follow-up period
  CFB of vital signs to subsequent visits
The safety endpoints are listed below for both phase I and IIa portions | from visit 2 to 12-month follow-up period
  CFB of AFP, CEA, CA199, SCC, IgA, anti-EBV, β-HCG, CA125, CA153, and PSA to Visit 6 (Phase I) or Visit 10 (Phase IIa)

OTHER OUTCOMES:
The exploratory endpoints are listed below for both phase I and IIa portions | from visit 2 to 12-month follow-up period
  Immunological markers, including CD3, CD4, CD8 surface markers, IgG, IgM, anti-HLA antibodies and Panel Reactive Antibody Assay in whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Woei C Shyu, Study Chair — Ever Supreme Bio Technology Co., Ltd.
Locations (1):
- China Medical University Hospital, Taichung, Non-US, Taiwan